CLINICAL TRIAL: NCT03917199
Title: Utility of Regadenoson Low-dose Dynamic Computed Tomography for Myocardial Perfusion Assesment (ULYSSES Study).
Acronym: ULYSSES
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2015/19/B/NZ5/03502
Record Dates: First submitted 2017-03-02; First posted 2019-04-16 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Myocardial Perfusion Imaging; Computed Tomography; Coronary Artery Disease
Keywords: myocardial perfusion imaging; computed tomography perfusion; regadenoson; dynamic perfusion; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The ULYSSES study is a single-center, prospective study aimed at evaluation of myocardial ischemia using regadenoson low-dose dynamic computed tomography myocardial perfusion imaging (CTP) in patients diagnosed with intermediate coronary artery stenoses in referrence to the magnetic resonance myocardial perfusion imaging (MR MPI).

DETAILED DESCRIPTION:
The ULYSSES study is a single-center, prospective study aimed at evaluation of myocardial ischemia using regadenoson low-dose dynamic computed tomography myocardial perfusion (CTP) in patients diagnosed with intermediate coronary artery stenoses in referrence to the magnetic resonance myocardial perfusion imaging (MR MPI).

The main objectives of the study are:

* to evaluate feasibility of low - dose regadenoson dynamic computed tomography myocardial imaging protocol
* to assess the diagnostic value of quantitative dynamic CTP based absolute parameters (myocardial blood flow - MBF, myocardial blood volume - MBV, perfused capillary blood volume - PCBV, peak value - PV, time to peak - TTP) in reference to magnetic resonance myocardial perfusion imaging
* to assess the diagnostic value of quantitative dynamic CTP based relative parameters (relative myocardial blood flow - MBFR, relative myocardial blood volume - MBVR, relative perfused capillary blood volume - PCBVR, relative peak value - PVR, relative time to peak - TTPR) in reference to magnetic resonance myocardial perfusion imaging
* evaluation of safety of regadenoson low-dose dynamic CTP.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* signing written, informed consent by the patient for participation in the study
* patients who are asymptomatic or with symptoms of stable coronary heart disease
* intermediate coronary artery stenosis of at least one coronary artery in CTCA

Exclusion Criteria:

* the symptoms of unstable ischemic heart disease and /or myocardial infarction,
* the history of myocardial infarction
* patients with impaired renal function (GFR <60 mL)
* contraindications for computed tomography or magnetic resonance imaging (including pregnancy, the presence of a cardiac pacemaker or cardioverter-defibrillator, claustrophobia, the presence of metal elements, etc.);
* contraindications to the administration of iodine contrast media (including allergy to contrast, unstable hyperthyroidism, etc.)
* contraindications to administration of regadenosone (hypersensitivity to the active substance, second or third degree atrioventricular block or other sinus node dysfunction, unstable angina, hypotension, decompensated heart failure, etc.);
* heart failure with impaired left ventricular systolic function
* a significant valvular heart disease
* presence of aortic aneurysm or aortic dissection
* persistent atrial fibrillation / atrial flutter
* hypertrophic cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population as described in inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-11; Primary Completion 2019-07 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of feasibility of regadenoson low - dose dynamic computed tomography perfusion protocol. | 24 months
  Evaluation of the quality of CTP images asessed by experienced readers.
Assessment of ischemia in regadenoson low-dose dynamic CTP in reference to magnetic resonance myocardial perfusion imaging (MR MPI). | 24 months
  The presence of ischemia in CTP per myocardial segment.

OTHER OUTCOMES:
Evaluation of radiation dose during regadenoson low-dose dynamic CTP. | 24 months
  Assessment of DLP (dose lenght product).
Evaluation of contrast agent dose during regadenoson low-dose dynamic CTP. | 24 months
  Assessment of contast agent dose (ml).

CONTACTS AND LOCATIONS:
Overall Officials: Cezary Kepka, MD, PhD, Principal Investigator — Institute of Cardiology, warsaw, PL
Locations (1):
- Institute of Cardiology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No